CLINICAL TRIAL: NCT05777291
Title: IntelligentCare: the Impact of a Wearable-based Intervention in an Ambulatory Hospital Setting to Improve Health in Multimorbidity Through Physical Activity and Sleep
Brief Title: IntelligentCare: Wearable-based Intervention
Acronym: ICare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GLSMED Learning Health S.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 500
Record Dates: First submitted 2023-03-03; First posted 2023-03-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Multimorbidity; Exercise; Sleep
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: unblinded randomized trial with blinded outcome assessors
Who Masked: Outcomes Assessor
Masking Description: The masking procedure will involve blinding the outcome assessors to the treatment allocation of the patients. This means that the outcome assessors will be kept unaware of whether the patients are wearing the device or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Patients will be given physical activity recommendations ABD will be using the study devices: activity watch (Fitbit Sense) and a sleep monitoring mattress (Withings, Sleep Analyzer)
  Interventions: Device: Activity watch monitoring; Device: Sleep mattress monitoring; Behavioral: Physical activity counseling
- Control arm (Active Comparator): Patients will be given physical activity recommendations only
  Interventions: Behavioral: Physical activity counseling

INTERVENTIONS:
Device: Activity watch monitoring — Patients will be using activity devices during the study period
  Arms: Experimental arm
Device: Sleep mattress monitoring — Patients will be using sleep mattress during the study period
  Arms: Experimental arm
Behavioral: Physical activity counseling — Physical activity counseling in accordance to the Swedish model

SUMMARY:
The benefits of physical activity and adequate sleep are well documented, and their importance strengthens with the increasing prevalence of chronic diseases and multimorbidity. Interventions to promote physical activity and sleep that use commercial activity trackers may be useful non-pharmacological approaches to managing individual health; however, limited evidence exists on their use to improve physical activity in elderly patients with multimorbidity. This study aims to measure the effects of behavioral change techniques (BCTs) delivered by a wearable device on physical activity (PA) and quality of sleep (QS) in elderly patients with multimorbidity. The investigators designed an open-label randomized controlled trial with participants recruited through primary care and a specialist outpatient clinic. Participants must be more than 65 years old, have multimorbidity, and have access to smartphones. All eligible participants will receive PA promotion content and will be randomly assigned to wear a smartwatch. The primary outcome will be the participants' PA measurement at six months using the IPAQ-SF. Secondary outcomes will include changes in the participants' frailty status, biometric measurements, quality of life, and biopsychosocial assessments. A sample size of 40 participants per arm was calculated to detect group differences, with 50 participants recruited and randomized into each arm. This study aims to contribute to a better understanding of PA patterns and the impact of smartwatch-based PA interventions in patients with multimorbidity. The trial's findings are expected to improve our understanding of how physical activity patterns, patient-reported outcomes (PROMs), and healthcare resource utilization are linked in patients with multiple medical conditions. The study will use a registry for locally developed PROMs and data from the participants' medical records to determine how wearable data and medical information data can be used to predict PROMs and unplanned hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* Multimorbidity defined as the presence of two or more of the following chronic conditions: hypertension, depression or anxiety, chronic musculoskeletal conditions causing pain or limitation, arthritis and/or rheumatoid arthritis, osteoporosis, asthma, COPD, ischemic heart disease, peripheral artery disease, heart failure, cerebrovascular diseases, chronic stomach or colon conditions, chronic hepatitis, diabetes mellitus, thyroid disorders, any active cancer in the previous five years, chronic kidney disease, chronic urinary conditions, hyperlipidemia, and obesity
* Must have access to their smartphones

Exclusion Criteria:

* patients who are sufficiently physically active (IPAQ-SF > 150 min aerobic physical activity per week)
* existing absolute contraindication for PA according to the American College of Sports Medicine (acute myocardial infarction within two days, ongoing unstable angina, uncontrolled cardiac arrhythmia with hemodynamic compromise, active endocarditis, symptomatic severe aortic stenosis, decompensated heart failure, acute pulmonary embolism, pulmonary infarction, deep venous thrombosis, acute myocarditis or pericarditis, acute aortic dissection, physical disability that precludes safe and adequate testing)
* poor comprehension of Portuguese language
* disabling neurological disorder (defined as mRankin score ≥4), severe psychiatric illness, learning disability, dementia and cognitive impairment, registered blind
* housebound or resident in a nursing home or non-ambulant
* advanced cancer
* scheduled for surgery within five months after the first consultation
* orthopedic or rheumatologic diseases with severe impairment
* chronic pain syndromes with inherently reduced mobility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 6 months after study entry
  Physical activity measured trough International Physical Activity Questionnaire Short Form. The responses to these questions are used to calculate an individual's total physical activity level, expressed in metabolic equivalent of task (MET) minutes per week. The IPAQ-Sf assigns a MET value to each activity reported by the individual and multiplies this value by the reported duration of the activity to calculate the total MET-minutes per week for each domain. The total MET-minutes per week for all domains are then summed to give the total physical activity level for the individual. The results of the IPAQ-Sf can be used to classify individuals into different categories of physical activity levels, such as low, moderate, or high.

SECONDARY OUTCOMES:
Physical performance | 6 months after study entry
  Assessed trough Short Physical Performance Battery. It is a non-invasive test designed to assess physical performance in older adults, with three parts. Each component of the SPPB test is scored on a scale of 0 to 4 points, with a maximum total score of 12 points. A higher score indicates better physical performance and mobility.
Fall risk | 6 months after study entry
  Assessed trough a validated 4-question questionnaire where any positive question indicates fall risk. More positive answers indicate greater risk.
Weight | 6 months after study entry
  Weight measured in Kgs and reported in isolation and with Body Mass Index
Abdominal circunference | 6 months after study entry
  Abdominal circunference in cm
Calf circunference | 6 months after study entry
  Calf circunference in cm
Health-related quality of life | 6 months after study entry
  Short Form Survey 12 that generates two summary scores, the physical component summary (PCS) score and the mental component summary (MCS) score. The PCS score reflects an individual's physical health status and the MCS score reflects their mental health status. Scores are standardized, with a mean of 50 and a standard deviation of 10, so scores above 50 indicate better health status than the reference population and scores below 50 indicate worse health status.
Biopsychosocial complexity and health care needs | 6 months after study entry
  INTERMED self-assessment questionnaire consists of 23 items that assess different aspects of a patient's health and social situation, such as the presence of chronic pain, mental health problems, social support, and functional impairment. Results are used to calculate an overall INTERMED score, which ranges from 0 to 60. The higher the score, the greater the complexity of the patient's health and social situation.
Unplanned hospital admissions | 6 months after study entry
  Number of emergency department visits and unplanned hospital admissions during study period

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Neves, MD, Principal Investigator — Researcher
Locations (1):
- Hospital da Luz Learning Health, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neves B, Haghighi ED, Pereira HV, Costa F, Carlos JS, Ferreira D, Moreno P, Ferreira PM, Machado J, Goncalves B, Moreira JM, Leite F, da Silva NA. Impact of a wearable-based physical activity and sleep intervention in multimorbidity patients: protocol for a randomized controlled trial. BMC Geriatr. 2023 Dec 14;23(1):853. doi: 10.1186/s12877-023-04511-y. PMID 38097933